CLINICAL TRIAL: NCT05877482
Title: Effect of Insoles With and Without Short Foot Exercises on Pain, Disability and Foot Posture in Children With Pes Planus
Brief Title: Pediatric Pes Planus: Effect of Insoles With and Without SFE
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Riphah International University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: REC/RCR & AHS/22/0719
Record Dates: First submitted 2023-05-18; First posted 2023-05-26 (Actual); Last update posted 2023-05-26 (Actual); Status verified 2023-05

CONDITIONS: Flexible Flatfoot
Keywords: Short foot exercises; Pes Planus; Flat Feet; Insoles; Foot Posture Index; Navicular drop test
MeSH Terms: conditions — Flatfoot | interventions — Foot Orthoses

STUDY DESIGN:
Who Masked: Participant, Investigator
Masking Description: Group assignment and short foot exercises training was conducted by the second physical therapist to provide blindness.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Experimental Group (Experimental): Short foot exercises with internal shoe modification (a medial longitudinal arch support) will be performed daily for six weeks.
  Interventions: Other: Short foot exercises; Other: Insoles
- Control Group (No Intervention): Only internal shoe modification will be performed by placing a medial longitudinal arch support insoles inside the shoe.

INTERVENTIONS:
Other: Short foot exercises — A total of 26 participants with pes planus were assigned to the short-foot exercises group (n = 13) and the control group (n = 13). Both groups will be informed about pes planus, usual foot care, and appropriate footwear with foot insoles. In experimental group Short foot exercises (SFE) and internal shoe modification will be performed by placing a medial longitudinal arch support insoles inside the shoe. Exercises will be performed daily for six weeks.
  Arms: Experimental Group
Other: Insoles — In control group only internal shoe modification will be performed by placing medial longitudinal arch support insoles inside the shoe. Group assignment and SFE training will be conducted by the second physical therapist to provide blindness.
  Arms: Experimental Group

SUMMARY:
The goal of this randomised control trial is to determine the effects of insoles with and without short foot exercises on pain, disability and foot posture in children with pes planus.

The main question[s] it aims to answer are:

1. What are the effects of insoles on pain, disability, and foot posture in children with pes planus?
2. What are the effects of short foot exercises on pain, disability, and foot posture in children with pes planus?
3. What are the combined effects of insoles and short foot exercises on pain, disability, and foot posture in children with pes planus?
4. Is there a significant difference between the effects of insoles alone versus insoles with short foot exercises on pain, disability, and foot posture in children with pes planus?

Participants will be asked to signed consent form and divided into two groups. Experimental group will be asked to performed short foot exercises with internal shoe modification (a medial longitudinal arch support) daily for six weeks and Control Group will be asked to perform only internal shoe modification by placing a medial longitudinal arch support insoles inside the shoe.

Researchers will compare:

1) Insoles only vs insoles + short foot exercises: This comparison would involve evaluating the effects of wearing insoles alone compared to wearing insoles and performing short foot exercises together to see effect on pain, disability, and foot posture among pes planus children between age group of 08 to 16 years.

DETAILED DESCRIPTION:
All participants will be informed about the study, and an informed consent form was signed by each participant. A total of 26 participants with pes planus will be assigned, to the short-foot exercises group (n = 13) and the control group (n = 13). Both groups will be informed about pes planus, usual foot care, and appropriate footwear with individually designed foot insoles. In experimental group Short foot exercises (SFE) and internal shoe modification will be performed by placing an individually designed medial longitudinal arch support insoles inside the shoe. Exercises will be performed daily for six weeks. While in control group only internal shoe modification will be performed. Short-foot exercises group will be performed the exercises daily for 6 weeks. Normality of data checked by the Shapiro wilk test. If the P-value is more than 0.05 then para metric test will applied and if P value is less than 0.05 than it is non-parametric. SPSS version 25.0 statistical software will be used. This study will examine the effects of individually designed insole in pes planus treatment with and without short foot exercises to improve the physical performance parameters and minimize the complaints of the individuals with pes planus.

ELIGIBILITY:
Inclusion Criteria:

* Having bilateral pes planus according to Navicular Drop (ND) exceeding 10 mm
* six item Foot Posture Index (FPI) score 6 to 12

Exclusion Criteria:

* Children having rigid pes planus,
* Hallux valgus,
* Hallux rigidus,
* Epin calcanei,
* Systemic, neurological or orthopedic problems that can affect the lower extremity,
* History of surgery on the lower extremities.
* Musculoskeletal pathologies, open wound in foot or a previous spinal/lower limb surgery

Ages: 8 Years to 16 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 26 (Estimated)
Dates: Start 2023-03-01 (Actual); Primary Completion 2023-08-01 (Estimated); Study Completion 2023-09-01 (Estimated)

PRIMARY OUTCOMES:
Navicular Drop (ND) test for inclusion criteria | 1st week
  The Navicular Drop Test (NDT) was first described by Brody in 1982 as a means of quantifying the amount of foot pronation in runners. It is the one of the static foot assessment tool and is intended to represent the sagittal plane displacement of the navicular tuberosity from a neutral position i.e. Subtalar joint neutral to a relaxed position in standing.

SECONDARY OUTCOMES:
Six item Foot Posture Index (FPI) | 6th week
  The FPI-6 is a novel method of rating foot posture using set criteria and a simple scale. It is a clinical tool used to quantify the degree to which a foot is pronated, neutral or supinated. It is a measure of standing foot posture and so is not a replacement for gait assessment where time and facilities exist. It is however a more valid approach than many of the static weight bearing and non-weight bearing goniometric measures currently used in clinic.
Pain and disability were assessed by pain and disability subscales (both include 9 items) of the Foot Function Index (FFI) | 6th week
  A Foot Function Index (FFI) was developed in 1991 to measure the impact of foot pathology on function in terms of pain, disability and activity restriction. [1] It is a self-administered index consisting of 23 items divided into 3 sub-scales. Both total and sub-scale scores are produced.

CONTACTS AND LOCATIONS:
Overall Officials: Dr. Arnab Altaf, BSPT,Mphil, Principal Investigator — Riphah International University
Locations (1):
- Children Hospital Lahore, Lahore, Punjab Province, Pakistan

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Alazzawi S, Sukeik M, King D, Vemulapalli K. Foot and ankle history and clinical examination: A guide to everyday practice. World J Orthop. 2017 Jan 18;8(1):21-29. doi: 10.5312/wjo.v8.i1.21. eCollection 2017 Jan 18. PMID 28144575
- [Background] Gwani AS, Asari MA, Mohd Ismail ZI. How the three arches of the foot intercorrelate. Folia Morphol (Warsz). 2017;76(4):682-688. doi: 10.5603/FM.a2017.0049. Epub 2017 May 29. PMID 28553850
- [Background] Acak M. The effects of individually designed insoles on pes planus treatment. Sci Rep. 2020 Nov 12;10(1):19715. doi: 10.1038/s41598-020-76767-y. PMID 33184442
- [Background] Caravaggi P, Pataky T, Gunther M, Savage R, Crompton R. Dynamics of longitudinal arch support in relation to walking speed: contribution of the plantar aponeurosis. J Anat. 2010 Sep;217(3):254-61. doi: 10.1111/j.1469-7580.2010.01261.x. Epub 2010 Jul 14. PMID 20646107
- [Background] Hashimoto T, Sakuraba K. Strength training for the intrinsic flexor muscles of the foot: effects on muscle strength, the foot arch, and dynamic parameters before and after the training. J Phys Ther Sci. 2014 Mar;26(3):373-6. doi: 10.1589/jpts.26.373. Epub 2014 Mar 25. PMID 24707086
- [Background] McCormack AP, Ching RP, Sangeorzan BJ. Biomechanics of procedures used in adult flatfoot deformity. Foot Ankle Clin. 2001 Mar;6(1):15-23, v. doi: 10.1016/s1083-7515(03)00072-x. PMID 11385922
- [Background] Chevalier TL, Chockalingam N. Effects of foot orthoses: How important is the practitioner? Gait Posture. 2012 Mar;35(3):383-8. doi: 10.1016/j.gaitpost.2011.10.356. Epub 2011 Nov 21. PMID 22104292
- [Background] Nawoczenski DA, Saltzman CL, Cook TM. The effect of foot structure on the three-dimensional kinematic coupling behavior of the leg and rear foot. Phys Ther. 1998 Apr;78(4):404-16. doi: 10.1093/ptj/78.4.404. PMID 9555923
- [Background] Yurt Y, Sener G, Yakut Y. The effect of different foot orthoses on pain and health related quality of life in painful flexible flat foot: a randomized controlled trial. Eur J Phys Rehabil Med. 2019 Feb;55(1):95-102. doi: 10.23736/S1973-9087.18.05108-0. Epub 2018 Mar 16. PMID 29553223
- [Background] Unver B, Erdem EU, Akbas E. Effects of Short-Foot Exercises on Foot Posture, Pain, Disability, and Plantar Pressure in Pes Planus. J Sport Rehabil. 2019 Oct 18;29(4):436-440. doi: 10.1123/jsr.2018-0363. Print 2020 May 1. PMID 30860412
- [Background] Yildirim Sahan T, Aydogan Arslan S, Demirci C, Oktas B, Sertel M. Comparison Of Short-Term Effects Of Virtual Reality and Short Foot Exercises In Pes Planus. Foot (Edinb). 2021 Jun;47:101778. doi: 10.1016/j.foot.2021.101778. Epub 2021 Jan 21. PMID 33962115
- [Background] Taspinar O, Kabayel DD, Ozdemir F, Tuna H, Keskin Y, Mercimek OB, Sut N, Yavuz S, Tuna F. Comparing the efficacy of exercise, internal and external shoe modification in pes planus: A clinical and pedobarographic study. J Back Musculoskelet Rehabil. 2017;30(2):255-263. doi: 10.3233/BMR-150399. PMID 27858680